CLINICAL TRIAL: NCT04752423
Title: Assessment of Patient Preoperative Anxiety by Nurse Anesthetist
Brief Title: Nurse Anesthesist Assessment of Patient Preoperative Anxiety
Acronym: EVALANXI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: EPP/2020/01
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Anxiety; Anesthesia, General
Keywords: Preoperative anxiety; Concordance; Self-assessment assessment of anxiety; Nurse anesthesist hetero-assessment of anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PATIENT group: Adult patients shedule for general anesthesia
  Interventions: Other: Pre operative assessment
- NURSE group: Nurse anesthesist in charge of the corresponding patient
  Interventions: Other: Pre operative assessment

INTERVENTIONS:
Other: Pre operative assessment — Anxiety assessment : Numeric rating scale (patient and caregiver), APAIS scale (patient), Covi Scale (Caregiver)
  Verbalization : anesthesia-related concerns (expressed by patient and considered by caregiver)

SUMMARY:
Preoperative anxiety is a major concern for patients who undergo surgery. To accurately identify anxious patient is therefore crucial to improve perioperative patient care. Preoperative anxiety remain highly difficult to quantify in current practice. Many patient fail to express their anxiety and the assessment of the level of anxiety is mainly based on heteroevaluation by caregivers. Nurse anesthetists provide closed support to patient prior to the induction of anesthesia. The aim of the study is to assess whether nurse anesthetist accurately assess patient preoperative anxiety from arrival to the operating room to the induction of anesthesia.

DETAILED DESCRIPTION:
EVALANXI is a single-center prospective observational study. The main objective of the study is to assess whether the assessment of preoperative anxiety by nurse anesthetist (hetero-assessment) accurately estimate the level of anxiety reported by the patient from arrival to the operating room to the induction of anesthesia (self-assessment).

ELIGIBILITY:
Patient Inclusion Criteria:

* Age > 18 years old
* Patients with ASA 1, ASA 2 ou ASA 3
* Patients undergoing planned surgery with general anesthesia

Patient Exclusion Criteria:

* Age <18
* Refusal, inability to oral consent
* Cardio-thoracic surgery or emergency surgery
* Patient with dementia, medically diagnosed psychiatric disorder, inability to answer questions

Nurse anesthetist Inclusion Criteria:

* Nurse anesthesis in charge of the corresponding patient

Nurse anesthetist Exclusion Criteria:

* Assessment of the preoperative anxiety of a previously included patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient undergoing general anesthesia and the corresponding nurse anesthetist in charge of the patient.
  To avoid any learning effect, each nurse can only participate once in the study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Comparison of preoperative anxiety level expressed by the patient (self-assessment) with that estimated by murse anesthetist (hetero-assessment) | Self- and hetero-assessment will be performed peroperatively during the period from arrival in the operating room to the induction of general anesthesia.
  Agreement between patient's Numeric Rating Scale (NRS from 0 to 10) and nurse anesthetist NRS (kappa coefficient)

SECONDARY OUTCOMES:
Patient anxiety self assessment : NRS (from 0 to 10) versus Amsterdam Preoperative Anxiety and Information (APAIS) scale (from 6 to 30) | Self- and hetero-assessment will be performed preoperatively during the period from arrival in the operating room to induction of general anesthesia.
  correlation between NRS and APAIS scale
Patient's Anxiety assessment by caregiver : NRS (from 0 to 10) versus Covi scale from 3 to 15) (Lipman & Covi 1976) | Self- and hetero-assessment will be performed preoperatively during the period from arrival in the operating room to induction of general anesthesia.
  correlation between NRS and Covi scale
Reliability of hetero-assessment performed by caregiver | Hetero-assessment will be performed preoperatively during the period from arrival in the operating room to induction of general anesthesia.
  sub group analysis based on nurse anesthetist professional experience
Anesthesia-related concerns | Anesthesia-related concerns observed by the patient and the corresponding nurse anesthetist will be collected preoperatively from arrival in the operating room to induction of general anesthesia.
  Comparison between the patient's expression and caregiver's estimate

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided